CLINICAL TRIAL: NCT07373587
Title: Preventing Hospital Associated Disability in Older Patients: Individualized Nutrition and Exercise Strategy, a Randomized Controlled Trial
Brief Title: Preventing Hospital Associated Disability in Older Patients: Individualized Nutrition and Exercise Strategy
Acronym: PrevHAD RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Suetta, Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: p-2026-20660; 3165-00244B (Other Grant/Funding Number: Independent Research Fund Denmark)
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Sarcopenia in Elderly; Hospital Associated Disability; Malnutrition Elderly; Physical Function
Keywords: Older; Hospitalized; Sarcopenia; Malnutrition; Exercise intervention
MeSH Terms: conditions — Sarcopenia; Malnutrition | interventions — Exercise

STUDY DESIGN:
Masking Description: Outcomes at discharge will be measured by a different investigator than at baseline, to mask the baseline measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will recieve usual care at the geriatric care unit, with mobility exercise performed based on individual preferences and ability, performed by regular care personelle and regular physiotherapy staff.
- Exercise intervention (Experimental): The exercise intervention group will recieve two times 30 minutes of supervised exercise (mobility and resistance exercise) every day during their stay at the geriatrich care unit.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The participants in the intervention group will recieve supervised exercise two times 30 minutes each day during hospitalization. The first exercise pass consists of resistance exercise, and can be performed supine in bed, sitting on the edge of the bed, and in a close-by exercise area, based on participants mobility level. The second exercise pass consists of mobility exercise, aiming to transfer the participant from supine in the bed to sitting position, transfer to chair, walking with or without walking aids or walking on stairs.
  Other Names: Training; Physiotheraphy
  Arms: Exercise intervention

SUMMARY:
Aproximately a third of persons older than 70 years lose physical function and ability to take care of themselves during a stay at a hospital. This is associated to an increased risk of readmission and mortality. Earlier research has shown that insufficient nutrition and physical activity during hospital stay, leading to a loss in muscle mass and strength, plays an important role in this fall in functionality. This study aims to examine if a structured and supervised resistance and mobility exercise intervention, can prevent this fall in functional ability during hospital stay among older patients. The Impact of nutritional status will be investigated by registrering caloric, protein and hydtrational intake during the study period.

DETAILED DESCRIPTION:
Older persons are highly susceptible to hospital associated disability (HAD), defined by a loss of physical function during hospitalization, leading to increased dependency, morbidity, and mortality. Key factors in developing HAD are physical inactivity, malnutrition and dehydration, leading to a decline in muscle mass and muscle strength. Therefore, there is a need to develop effective nutritional and exercise interventions for older patients, during hospitalization. Hypothesis: This study expects that a mobility-graded individualized exercise intervention will effectively prevent a decline in activities of daily living (ADL) function, mobility level, physical function, muscle and strength, and reduce the length of stay, risk of re-admission and mortality among older patients during hospital stay. The investigators furthermore hypothesize that sufficcient nutrition and hydration will improve the impact of the exercise intervention. The study is designed as a randomized controlled trial, and will include 360 participants, men and women, ≥ 65 years old from the geriatric care unit of Bispebjerg Hospital, Denmark. After inclusion, participants will have estimated nutritional status, frailty and mobility, muscle mass and strength, physical function, ADL function, cognitive function and quality of life. Futhermore, blood samples for analysis of anabolic and inflammatory biomarkers as well as microbiome samples will be taken at baseline testing. After baseline testing, the participants will be divided randomely 1:1 into a control group and an intervention group. All participants will have nutritional and hydrational intake registered and wear accelerometers during the study period. The participants in the intervention group will receive 2 x 30 minutes supervised exercise (resistance and mobility) every day during the stury period. At discharge or transfer from the geriatric care unit, participants will be tested for mobility, muscle mass and strength, physical function, ADL function, cognitive function and quality of life. 1 Month after discharge from hospital, the participants will recieve af telefon interview, reporting on ADL-function, mobility, quality of life and nutritional status. Participants succesfully reached by telephone interview, will be asked further permission for a homevisit, where muscle strength and mass, physical function, mobility, cognitive function and ADL function will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized at the geriatric ward
* Speak Danish or English
* Ability to give informed consent

Exclusion Criteria:

* Moderate to severe Dementia
* Manifest delirium

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2026-02-03 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Changes in activities of daily living (ADL) function, by Barthel index-100 | From enrollment to discharge/transfer from the geriatric care unit (aproximately 5 days), measured again 1 month after discharge.
  describes the level of independence in activities of daily living, score of 0 equals total dependence and a score of 100 equals total independence

SECONDARY OUTCOMES:
Changes in mobility by Cumulated Ambulation Score | From enrollment to discharge/transfer from the geriatric care unit (aproximately 5 days), measured again 1 month after discharge
  Cumulated Ambulation Score (assesed mobility, 0 (lowest)-6(highest))
Changes in Knee extension strength, | From enrollment to discharge/transfer from the geriatric care unit (aproximately 5 days), measured again 1 month after discharge.
  (Knee extension strength, maximal voluntary contraction, newton meter)
Changes in Hand Grip Strength | From enrollment to discharge/transfer from the geriatric care unit (aproximately 5 days), measured again 1 month after discharge.
  Hand grip strength, kilogram
Changes in Sit-to-stand performance | From enrollment to discharge/transfer from the geriatric care unit (aproximately 5 days), measured again 1 month after discharge.
  Sit-to-stand test, number of repetitions in 30 seconds, continous scale
Changes in Gait speed | From enrollment to discharge/transfer from the geriatric care unit (aproximately 5 days), measured again 1 month after discharge.
  Gait speed, velocity (meters/seconds)
Changes in Quadriceps muscle thickness | From enrollment to discharge/transfer from the geriatric care unit (aproximately 5 days), measured again 1 month after discharge.
  Quadriceps muscle thickness, ultrasound, millimeters
Changes in muscle mass | From enrollment to discharge/transfer from the geriatric care unit (aproximately 5 days), measured again 1 month after discharge.
  muscle mass, bioimpedance analysis, kilogram
Changes in appetite | From enrollment to discharge/transfer from the geriatric care unit (aproximately 5 days), measured again 1 month after discharge.
  appetite, simplified nutritional appettite questionaire. Scale, 4-20, lower values indicates higher risk of insufficient nutritional intake
Changes in quality of life | From enrollment to discharge/transfer from the geriatric care unit (aproximately 5 days), measured again 1 month after discharge.
  quality of life, EuroQol- 5Dimensions-5 levels, questionaire, scale from 1-5 i each of five dimensions, higher scores indicates lower quality of life
Readmission 30 days from discharge | From inclusion to 30 days after discharge from hospital
  Participants readmitted to the hospital within 30 days of discharge, categorical yes or no
Mortality 30 days, 90 days and 1 year after discharge | From inclusion to 1 year after discharge from hospital
  Participant diseased at 30 days, 90 days or 1 year after discharge from hospital, categorical, yes/no
Changes in municipal care needs at discharge, 1 month and 3 months after discharge | Retrospectively 14 days berfore inclusion to 3 months after discharge from hospital
  Need for municipal care services, number of weekly visits, minutes of care service
Discharge destination | From inclusion to discharge from hospital (aproximately 5 days after inclusion)
  Discharged to own home, temporary rehabillitation or permanent care facility, categorical, yes or no
Physical activity during hospitalization | From inclusion to discharge from hospital (aproximately 5 days after inclusion)
  Steps taken and time upright, accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Suetta, Professor, Principal Investigator — Geriatric research unit, Bispebjerg hospital, Copenhagen
Locations (1):
- Bispebjerg Hospital, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
We will share the protocol for the exercise intervention, as well as participants charecteristics and outcome data, in a data repository, when the data can be fully anonymized
Supporting Information: Study Protocol, SAP
Time Frame: When the main study is published, estimated 1. march 2028, with no end date
Access Criteria: Data repository, URL link within the published study